CLINICAL TRIAL: NCT05276882
Title: Improved Rehabilitation After Surgery and Hypnosis: Benefits Potentiated by a Preoperative Consultation
Acronym: RACHYP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-AOI-08
Record Dates: First submitted 2022-02-17; First posted 2022-03-11 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Gynecological Disease
Keywords: laparoscopic gynecological surgery
MeSH Terms: conditions — Genital Diseases, Female | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypnosis (Experimental)
  Interventions: Other: Hypnosis
- pre-surgery consultation (Active Comparator)
  Interventions: Other: pre-surgery consultation

INTERVENTIONS:
Other: Hypnosis — It will be an individualized hypnosis session of Ericksonian type. It consists in going through 3 phases: induction, dissociation, suggestion.
  The principle is to focus the patient's attention by talking to her or by surprising her, or by making her do an incongruous gesture which will make her focus on a restricted idea. She will reduce her field of consciousness and concentrate. This is where her work will begin, allowing her unconscious to function in order to find her solutions. At this moment, she is particularly receptive to suggestions and the hypnotherapist accompanies and guides her thoughts and her associations of ideas on therapeutic paths. He provokes a unique personal work which aims to promote healing.
  Arms: hypnosis
Other: pre-surgery consultation — Dialogue with the patient to clarify her expectations.
  * Answers to the patient's questions
  * Precision on the organization of the hospitalization if necessary
  * Information on the postoperative period with postural advice to facilitate the first getting up with less discomfort, and postures promoting rest in the postoperative period
  * Information on relaxation techniques and their interest (abdominal breathing)
  Arms: pre-surgery consultation

SUMMARY:
Today, patient management in the context of scheduled surgery must meet new requirements. The understanding of surgical aggression, the evolution of anesthesia and surgery techniques have allowed the birth of the protocol of Improved Rehabilitation After Surgery. The objective is a pain-free surgery, with a minimum of risks, with a global management of the patient and an active participation.

In 2019, the Nice University Hospital developed this program. Other non-medicinal techniques could promote the evolution of this program such as integrative medicine with, in this study case, hypnosis. Since 2002, thanks to its widely recognized effectiveness in the treatment of pain and in helping with care, its use has developed. A hypnosis session, proposed in the preoperative period, would considerably reduce the patient's anxiety, postoperative pain, a better and faster recovery with an easier healing: objectives of the Improved Rehabilitation After Surgery program. The patient's satisfaction would also be improved thanks to his active participation, in a greater comfort, which the investigators want to demonstrate by our work.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age ≥ 18 years
* Indication for laparoscopic gynecological surgery eligible for the Improved Rehabilitation After Surgery protocol
* Understanding of French essential
* Signature of informed consent
* Affiliation to a Social Security system

Exclusion Criteria:

* Patient with a history of psychiatric pathologies (Schizophrenia, Psychosis, Bipolarity)
* Deafness, intellectual deficiency not allowing comprehension
* Pregnant or breastfeeding women
* Women of childbearing age who are not using an effective method of contraception (pill, intrauterine device, vaginal ring, contraceptive skin patch, subcutaneous hormonal implant, surgical sterilization)
* Patient under guardianship or deprived of liberty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 55 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Patient anxiety | Up to 2 months
  Evolution of the patient's anxiety between the initial consultation and the day of the surgery.
  Anxiety will be measured using the Spielberger State Trait Anxiety Inventory (S.T.A.I.) To obtain the state-anxiety score, the scores obtained for the 20 items corresponding to the state-anxiety (items 1 to 20) are added together. If two or more items are not answered, the questionnaire cannot be used.
  The mean score for women in non-anxiety situations was 47.13 with a standard deviation of 10. A score higher than this indicates an anxious state.
  Very high score > 65 High score = 56 to 65 Average score= 46 to 55 Low score=36 to 45 Very low score < or = 35

SECONDARY OUTCOMES:
Patient satisfaction | day of discharge from hospital, average of 7 days
  Patient satisfaction will be assessed using the Enhanced Rehabilitation After Surgery protocol satisfaction questionnaire The questionnaire is composed of 9 questions exploring the patient's general feeling about her care, the clarity of the information received, pain, the Enhanced Rehabilitation After Surgery protocol
length of stay in hospital | the day of discharge from hospital, average of 7 days
  length of stay in hospital defined as the number of days between the day of surgery and discharge
use of injectable analgesic | Day 7 of the surgery
  Comparison of the number of patients having had an injectable analgesic prescription between Day 1 and Day 7 of the surgery (binary yes/no criterion).
  This evaluation is only relevant from Day 1 onwards, because at Day 0 it is very common to have to resort to parenteral analgesia.
speed of cicatrization | Day 7 of the discharge from hospital
  The speed of cicatrization will be evaluated in the postoperative period by means of the patient's logbook, which evaluates the evolution of the wound from day 2.
  The wound will be considered healed as soon as the patient answers that the dressing is clean.

CONTACTS AND LOCATIONS:
Overall Officials: Claire KOCIALKOWSKI, Principal Investigator — Nice University Hospital
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No